CLINICAL TRIAL: NCT00885781
Title: Clinical Study Comparing Safety and Efficacy of SMOFlipid, the New Generation Fat Emulsion, in Comparison With the Current Fat Emulsion Lipovenoes MCT at the Hospital
Brief Title: Efficacy and Safety Comparison Between SMOFlipid and Lipovenoes MCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 200803090M; SMOF-002-I P4
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-05

CONDITIONS: Gastrectomy; Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMOFlipid (Experimental)
  Interventions: Drug: lipid emulsion for TPN
- Lipovenoes MCT (Active Comparator)
  Interventions: Drug: lipid emulsion for TPN

INTERVENTIONS:
Drug: lipid emulsion for TPN — 1-2 g lipid emulsion /kgBW-day, for consecutive 5 days
  Other Names: SMOFlipid 20%

SUMMARY:
Comparison of efficacy and safety of two lipid emulsion products will be performed on gastrectomy patients postsurgically.

DETAILED DESCRIPTION:
The comparison of two lipid emulsion product will be performed. Patients who plan to accept gastrectomy will be consider for trial and signed content will be obtained. If the patient needs total parenteral nutrition (TPN) treatment after surgery for at least 5 days and meets all criteria, then he/she will be enrolled and randomized to ether of the groups, SMOFlipid or Lipovenoes MCT. During the treatment period, efficacy variables and safety variables will be measured. Life quality evaluation will also be performed through questionnaires collection.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 ~ 75 years old
2. Postoperative (gastrectomy) patients required parental nutrition for at least 5 days
3. Signed informed consent form

Exclusion Criteria:

1. Known hypersensitivity to fish-, egg- or soy protein or to any of the active substances or excipients
2. Known type IV hyperlipidemia, disturbances in lipid metabolism or hypertriglyceridemia. If the fasting S-triglyceride value at the time of inclusion is >2.26 mmol/l (>200 mg/dl) the subject must not be included
3. Severe liver insufficiency (total serum bilirubin ≧ 3 mg/dL or parental nutrition as a contraindication.)
4. Severe renal insufficiency with need for dialysis, chronic stable renal insufficiency defined as S-creatinine value of >3mg/dL (250 µmol/l), or dialysis/hemofiltration therapy
5. Over weight (BMI> 30kg/m2)
6. Severe blood coagulation disorders
7. Inborn abnormality in amino acid metabolism
8. Unstable conditions (e.g. severe post-traumatic conditions, uncompensated diabetes mellitus, acute myocardial infarction, stroke, embolism, metabolic acidosis, severe sepsis and hypotonic dehydration)
9. Known diabetic ketoacidosis 7 days prior to randomization.
10. Acute shock
11. General contraindications to infusion therapy: acute pulmonary oedema, hyperhydration, decompensated cardiac insufficiency
12. Pregnancy or lactation
13. Chemotherapy within 7 days before start of the trial
14. Participation in another clinical study with an investigational drug or an investigational medical device within 1 month prior to start of study or during the study
15. Already accept parental nutrition therapy.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-11; Primary Completion 2009-04 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Evidence for immunoregulatory effect of lipid emulsion products. | 1-5 days after treatment provided

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Tsan Lin, Dr., Principal Investigator — Chief of General Suery department
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan